CLINICAL TRIAL: NCT03134833
Title: Engaging Seronegative Youth to Optimize HIV Prevention Continuum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Tulane University Health Sciences Center (Other); University of California, San Francisco (Other); Friends Research Institute, Inc. (Other)
Responsible Party: Principal Investigator, Dallas Swendeman, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: U19HD089886 - Study 3; U19HD089886 (NIH)
Record Dates: First submitted 2017-04-04; First posted 2017-05-01 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: HIV; Mental Health; Substance Use; STI
Keywords: HIV; STI; Mental Health; Substance Use; Peer Support
MeSH Terms: conditions — Psychological Well-Being; Substance-Related Disorders; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Automated Messaging & Monitoring (Experimental): Youth randomized to the Automated Messaging and Monitoring Intervention (AMMI) arm will receive daily texts to motivate, inform, and refer youth to health care and HIV services. Message banks will focus on the HIV Prevention Continuum, with libraries of text messages dedicated to healthcare, wellness, sexual health, drug use and medication reminders (e.g., for PrEP) for young men-who-have-sex-with-men (MSM) and non-MSM.
  Youth will also receive a weekly monitoring survey that covers seven domains, including: use of PrEP/PEP, condomless sex, potential symptoms of acute HIV infection, potential symptoms of STI, excessive use of alcohol and/or drugs, feelings of sadness or depression, and housing or food insecurity.
  Interventions: Behavioral: Automated Messaging & Monitoring
- Peer Support (Experimental): Youth randomized to the Peer Support arm will be enrolled in private, online peer support groups, where they can post information and have discussions with other participants, guided broadly by topics relevant to the HIV Prevention Continuum. Peer Supporters will post to encourage and broadly guide discussion, while Coaches and Project Coordinators will be available to provide factual information (as needed), and remove inappropriate content. All youth will also receive AMMI messages.
  Interventions: Behavioral: Automated Messaging & Monitoring; Behavioral: Peer Support
- Coaching (Experimental): Youth randomized to the Coaching arm will have access to a dedicated Coach for crisis management, problem-solving, linkage to HIV and related services, and care coordination. The Coach's primary means of contact with youth will be electronic - using e-mail, social media, text messages - and phone calls. In person contacts may also occur. AMMI is also provided to all youth.
  Interventions: Behavioral: Automated Messaging & Monitoring; Behavioral: Coaching
- Coaching + Peer Support (Experimental): Youth randomized to the Coach + Peer Support arm will be enrolled in online, private peer support groups and have access to a Coach. As well as AMMI messages.
  Interventions: Behavioral: Automated Messaging & Monitoring; Behavioral: Peer Support; Behavioral: Coaching

INTERVENTIONS:
Behavioral: Automated Messaging & Monitoring — Youth will receive messages 1-5 messages per day for 24 months. Message banks of about 750 text messages (70-120/domain) will focus on the HIV Prevention Continuum, with messages dedicated to healthcare, wellness, sexual health, drug use and medication reminders (e.g., for PrEP) for MSM and non-MSM. Youth will be able to choose the time that they receive daily texts. Text timing and the frequency of texts (e.g., if the youth "comes out") will be updated at 4-month intervals.
  Youth will complete weekly monitoring surveys by text message. The survey will cover seven domains related to the HIV Prevention Continuum. In case of non-response, reminder messages will be sent to the youth. After three days of non-response, a follow-telephone call will occur.
Behavioral: Peer Support — Youth will be enrolled in online, private discussion groups.
  Peer Support will be offered by fellow participants and/or Youth Advisory Board members that have been trained in basic information on HIV, STI, drug use, mental health, homelessness, and stigma; using social media to create wall posts and use chat functions; and, how to initiate conversations on sensitive topics. By posting and responding to messages, Peer Supporters will encourage and broadly guide conversation related to the HIV Prevention Continuum, and other relevant topics.
  Coaches and Project Coordinators will be available to provide factual information (as needed), and remove inappropriate content.
  Arms: Coaching + Peer Support; Peer Support
Behavioral: Coaching — Youth will have access to a dedicated Coach to assist with crisis support and problem-solving, linkage to HIV and related services (e.g., for substance use, mental health), and care coordination. Coaches will be accessible electronically (using social media, e-mail, text messaging) and by phone. In cases where virtual support has failed, Coaches will be available in-person (e.g., to accompany a participant to a doctor's appointment). We anticipate that Coaches will provide each youth with 10 hours of support, on average, per year.
  Arms: Coaching; Coaching + Peer Support

SUMMARY:
The focus of this study (Engaging Seronegative Youth to Optimize HIV Prevention Continuum) - will be to stop HIV-related risk acts and to encourage youth at high risk for HIV to adopt antiretroviral medications as treatment and prevention (either pre exposure prophylaxis (PrEP) or post exposure prophylaxis) among gay, bisexual and transgender and/or homeless youth with contact with the criminal justice system in the HIV epicenters of Los Angeles and New Orleans. A cohort of 1500 youth at the highest risk of seroconverting over 24 months will be identified. The goal will be to optimize the HIV Prevention Continuum over 24 months. The proposed randomized controlled trial (RCT) aims to compare youth outcomes when randomized to one of four automated and person-mediated social media delivered intervention conditions: 1) Automated Messaging and Monitoring Intervention (AMMI) only (n=900) consisting of daily motivational, instructional, and referral text-messaging (SMS), and brief, weekly SMS monitoring surveys of outcomes; 2) Peer Support through social media plus AMMI (n=200) via private online discussion boards; 3) Coaching plus AMMI (n=200) to provide service linkages, eligibility support, appointment coordination and follow-up, communication with healthcare providers, and brief motivational and strengths-based counseling for linkage and retention to prevention, mental health, and substance abuse services; and, 4) Coaching plus Peer Support and AMMI (n=200).

DETAILED DESCRIPTION:
Despite dramatic improvements in the biomedical treatments for both preventing and treating HIV infection, American adolescents are increasingly likely to become infected, are not using ARV for prevention or treatment, and are not learning they are HIV seropositive when they have become infected. America's HIV epidemic among youth has more than doubled in the last 15 years and now represents 26% of the epidemic. These youth are not found in every community - geography is destiny in HIV prevention (www.AIDSVu.com). YLH are concentrated along I-95 on the East Coast, in Southern cities, and West Coast. Given the distribution of emerging infections, we have chosen two HIV epicenters, Los Angeles (LA) and New Orleans, to test a strategy to identify, link to care, and intervene to prevent HIV. Even in those two areas, adolescent HIV will not be found in every neighborhood. In LA, six neighborhoods account for 80% of HIV cases in the County - reflecting the concentration of HIV within neighborhoods and settings. In each epicenter, the youth at highest risk of infection will be gay, bisexual, and transgendered youth (GBTY), especially those who are Black and Latino. Homeless youth will also be at highest risk: the last HIV seroprevalence study showed a 5.3% rate among homeless youth. Youth who are incarcerated are at higher risk of being in risk setting and will be targeted for recruitment to this study. Having a sexual orientation as GBTY is highly stigmatizing and youth are developmentally challenged about who, when, how, and what to disclose their sexual orientation of HIV status to their families and their peers. Unfortunately 42% of GBTY's parents eject their children when children disclose being GBTY resulting in 40% of homeless youth being GBTY. Homeless GBTY had a seroprevalence of 24.8% in 1989.

The sites that typically serve GBTY and High Risk Youth (HRY) (gay-identified CBO and homeless shelters) in HIV epicenters only provide HIV testing to about 10% of youth currently. To effectively stop HIV among youth, a more integrated strategy that tests for HIV and STIs repeatedly, links youth to care, and helps youth access all HIV prevention strategies, including Pre Exposure Prophylaxis (PrEP) and Post Exposure Prophylaxis (PEP), is needed. The proposed research will test such a strategy.

To eliminate HIV among youth, scalable, efficacious, and cost-effective strategies are needed to optimize the HIV Prevention Continuum of repeat testing, linkage to biomedical and behavioral prevention, and retention and adherence over time to PrEP, PEP, condom use and reduced number of partners. The HIV Prevention Continuum is a framework for guiding prevention efforts.

Advances in mobile and social media technologies have created opportunities to engage and intervene with large numbers of youth at relatively low costs, technologies that permeate their daily routines. This study will use two primary technology platforms: text-messaging and social media. Text-messaging, email, internet and social media use are nearly universal among youth, including homeless youth. Rates of mobile phone, smartphone, and internet usage increase with age, and nearly 90% of young adolescents (age 13-17) having a mobile phone. Texting is particularly important for adolescents; 90% of those with phones text, typically receiving and sending 30 texts each day. Similarly, over 90% of adolescents under age 18 go online daily, more than half several times a day, which is facilitated the three quarters with smartphones that are crossing the digital divide. African-American and Latino youth have higher rates of smartphone and internet use than White. All of these rates increase for adolescents 18 and over. Ownership, access, and use rates are similar for homeless youth, although with less frequency and some inconsistency. Much of this online activity is driven by social media, particularly via smartphones, with over 70% of adolescents under 18, for example, using Facebook and other applications (about half also use Instagram and Snapchat).

The interventions proposed in this study will use text-messaging and social media to engage "youth where they're at" in the digital environment as preferences and functions change. Importantly, mobile phones continue to receive text-messages even when data plans run out of credit to use apps' and mobile-web browsers or send text-messages. Therefore, the core component our technology strategy will be text-messaging in the Automated Messaging and Monitoring Intervention (AMMI) for all youth in the cohort. Social media will be used by Peer Supporters to engage and support their peers through online discussion boards while Coaches will engage through social media, text-messaging, and voice and video-chats (however most acceptable to individual youth), as well as in person contacts. Mobile and social media technology-based engagement, retention, prevention, and mobilization strategies are likely to be scalable. This study will test whether they are also efficacious and cost-effective.

Upon study launch in April 2017, decisions were made with the funder to provide three-site STI testing at baseline and every follow-up assessment. In December 2018, the funder changed priorities and reduced support for STI testing to rectal testing only at baseline, 12- and 24-month follow-up, unless the participant displays STI symptoms or requests testing at other follow-up assessments. The funder has also decided to terminate the intervention and follow-up assessments at 12 months, rather than 24 months, for youth who are at lower behavioral risk for HIV acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Youth aged 12-24
* HIV-negative status
* Able to provide informed consent
* At high-risk* of HIV

  * Youth will be considered at high-risk of HIV based on their responses to a screening questionnaire, which assesses - HIV status; PrEP / PEP use; gender; race/ethnicity; sexual orientation; homelessness; history of probation/incarceration; history of hospitalization for mental health issues; history of substance abuse use and treatment; and, history of STI.

Exclusion Criteria:

* Youth under 12 years of age or above 24 years of age
* HIV-positive (if you become HIV-positive, they will be invited to participate in another, related ATN study)
* Unable to understand the study procedures due to intoxication or cognitive difficulties (any youth who appear to be under the influence of alcohol or drugs will be unable to enroll in the study but invited to return at a later date)
* Unable to provide voluntary written informed consent
* Do not meet aforementioned criteria for being at high-risk of HIV

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1478 (Actual)
Dates: Start 2017-05-06 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
HIV Testing | 24 months
  Self-reported # of times - lifetime, past 4 months (reported at four-month assessment points)
STI Testing | 24 months
  Self-reported # of times - lifetime, past 4 months (reported at four-month assessment points)
Condom Use Frequency | 24 months
  Self-reported condomless sex - lifetime, past four months - using Likert-type scale (reported on weekly surveys, at four-month assessment points)
PEP Use / Adherence | 24 months
  Self-reported current use, lifetime use, adherence, willingness to use - using Likert-type scale (all reported at four-month assessment points, adherence also reported on weekly surveys)
PrEP Use / Adherence | 24 months
  Self-reported current use, lifetime use, adherence; using Likert-type scale (all reported at four-month assessment points, adherence also reported on weekly surveys)
Sexual Partners | 24 months
  Self-reported # of sexual partners, # of female/male/transgender sexual partners - lifetime, past 4 months (reported at four-month assessment points)

SECONDARY OUTCOMES:
Mental Health Symptoms | 24 months
  Self-reported symptoms of anxiety and depression (reported on weekly surveys, at four-month assessment points)
Substance Use | 24 months
  Rapid Diagnostic Tests (RDTs) for alcohol, marijuana, methamphetamines, opiates, cocaine (at four-month assessment points); self-reported AUDIT-C measure (at four-month assessment points); self-reported excessive substance use (reported on weekly surveys)
Housing Insecurity | 24 months
  Self-reported housing insecurity (reported on weekly surveys, at four-month assessment points)

CONTACTS AND LOCATIONS:
Overall Officials: Dallas Swendeman, PhD, MPH, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Tulane University Health Sciences Center, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lightfoot M, Rotheram-Borus MJ. Interventions for high-risk youth. In: Peterson JL, DiClemente RJ, editors. Handbook of HIV prevention AIDS prevention and mental health. Dordrecht, Netherlands: Kluwer Academic Publishers; 2000. p. 129-45.
- [Background] Stricof RL, Kennedy JT, Nattell TC, Weisfuse IB, Novick LF. HIV seroprevalence in a facility for runaway and homeless adolescents. Am J Public Health. 1991 May;81 Suppl(Suppl):50-3. doi: 10.2105/ajph.81.suppl.50. PMID 2014885
- [Background] Swendeman D, Rotheram-Borus MJ, Comulada S, Weiss R, Ramos ME. Predictors of HIV-related stigma among young people living with HIV. Health Psychol. 2006 Jul;25(4):501-9. doi: 10.1037/0278-6133.25.4.501. PMID 16846325
- [Background] Adolescent sexual orientation. Paediatr Child Health. 2008 Sep;13(7):619-30. doi: 10.1093/pch/13.7.619. No abstract available. PMID 19436504
- [Background] Rotheram-Borus MJ, Fernandez MI. Sexual orientation and developmental challenges experienced by gay and lesbian youths. Suicide Life Threat Behav. 1995;25 Suppl:26-34; discussion 35-9. PMID 8553426
- [Background] D'Angelo LJ, Abdalian SE, Sarr M, Hoffman N, Belzer M; Adolescent Medicine HIV/AIDS Research Network. Disclosure of serostatus by HIV infected youth: the experience of the REACH study. Reaching for Excellence in Adolescent Care and Health. J Adolesc Health. 2001 Sep;29(3 Suppl):72-9. doi: 10.1016/s1054-139x(01)00285-3. PMID 11530306
- [Background] D'Augelli AR, Hershberger SL, Pilkington NW. Lesbian, gay, and bisexual youth and their families: disclosure of sexual orientation and its consequences. Am J Orthopsychiatry. 1998 Jul;68(3):361-71; discussion 372-5. doi: 10.1037/h0080345. PMID 9686289
- [Background] Durso LE, Gates GJ. Serving our youth: Finding from a national survey of service providers working with lesbian, gay, bisexual and transgender youth who are homeless or at risk of becoming homeless. Los Angeles: The Williams Institute with True Colors Fund and The Palette Fund; 2012.
- [Background] McNairy ML, El-Sadr WM. A paradigm shift: focus on the HIV prevention continuum. Clin Infect Dis. 2014 Jul;59 Suppl 1(Suppl 1):S12-5. doi: 10.1093/cid/ciu251. PMID 24926026
- [Background] International Advisory Panel on HIV Care Continuum Optimization. IAPAC Guidelines for Optimizing the HIV Care Continuum for Adults and Adolescents. J Int Assoc Provid AIDS Care. 2015 Nov-Dec;14 Suppl 1:S3-S34. doi: 10.1177/2325957415613442. Epub 2015 Nov 2. PMID 26527218
- [Background] Milburn NG, Liang LJ, Lee SJ, Rotheram-Borus MJ. Trajectories of risk behaviors and exiting homelessness among newly homeless adolescents. Vulnerable Child Youth Stud. 2009 Jan 1;4(4):346-352. doi: 10.1080/17450120902884068. PMID 21494426
- [Background] Ringwalt CL, Greene JM, Robertson MJ. Familial backgrounds and risk behaviors of youth with thrownaway experiences. J Adolesc. 1998 Jun;21(3):241-52. doi: 10.1006/jado.1998.0150. PMID 9657892
- [Background] Rosario M, Schrimshaw EW, Hunter J. Homelessness among lesbian, gay, and bisexual youth: implications for subsequent internalizing and externalizing symptoms. J Youth Adolesc. 2012 May;41(5):544-60. doi: 10.1007/s10964-011-9681-3. Epub 2011 Jun 7. PMID 21656284
- [Background] Dowshen N, Kuhns LM, Johnson A, Holoyda BJ, Garofalo R. Improving adherence to antiretroviral therapy for youth living with HIV/AIDS: a pilot study using personalized, interactive, daily text message reminders. J Med Internet Res. 2012 Apr 5;14(2):e51. doi: 10.2196/jmir.2015. PMID 22481246
- [Background] Rice E, Monro W, Barman-Adhikari A, Young SD. Internet use, social networking, and HIV/AIDS risk for homeless adolescents. J Adolesc Health. 2010 Dec;47(6):610-3. doi: 10.1016/j.jadohealth.2010.04.016. Epub 2010 Jun 23. PMID 21094441
- [Background] Rice E, Barman-Adhikari A. Internet and Social Media Use as a Resource Among Homeless Youth. J Comput Mediat Commun. 2014 Jan 1;19(2):232-247. doi: 10.1111/jcc4.12038. PMID 25328374
- [Background] Rotheram-Borus MJ, Tomlinson M, Gwegwe M, Comulada WS, Kaufman N, Keim M. Diabetes buddies: peer support through a mobile phone buddy system. Diabetes Educ. 2012 May-Jun;38(3):357-65. doi: 10.1177/0145721712444617. Epub 2012 Apr 30. PMID 22546740
- [Background] Swendeman D, Ramanathan N, Baetscher L, Medich M, Scheffler A, Comulada WS, Estrin D. Smartphone self-monitoring to support self-management among people living with HIV: perceived benefits and theory of change from a mixed-methods randomized pilot study. J Acquir Immune Defic Syndr. 2015 May 1;69 Suppl 1(0 1):S80-91. doi: 10.1097/QAI.0000000000000570. PMID 25867783
- [Background] Swendeman D, Ramanathan N, Comulada WS, Rotheram-Borus MJ, Estrin D. Efficacy of Daily Self- Monitoring of Health Behaviors and Quality of Life by Mobile Phone: Mixed-Methods Results from Two Studies with Diverse Populations. Annals of Behavioral Medicine. 2014;47:S263-S.
- [Background] Swendeman D, Rotheram-Borus MJ. Innovation in sexually transmitted disease and HIV prevention: internet and mobile phone delivery vehicles for global diffusion. Curr Opin Psychiatry. 2010 Mar;23(2):139-44. doi: 10.1097/YCO.0b013e328336656a. PMID 20087189
- [Background] Tomlinson M, Rotheram-Borus MJ, Doherty T, Swendeman D, Tsai AC, Ijumba P, le Roux I, Jackson D, Stewart J, Friedman A, Colvin M, Chopra M. Value of a mobile information system to improve quality of care by community health workers. S Afr J Inf Manag. 2013;15(1):10.4102/sajim.v15i1.528. doi: 10.4102/sajim.v15i1.528. PMID 25147730
- [Derived] Ma AM, Lewis KA, Wani M, Liu C, Ghalambor S, Yuva Raju R, Wong C, Swendeman D; ATN CARES Study Team; Abdalian SE, Arnold E, Bolan R, Bryson Y, Chaplin A, Comulada WS, Cortado R, Donahue C, Fernandez MI, Flynn R, Fournier J, Gertsch W, Ishimoto K, Jimenez S, Kerin T, Klausner J, Kussin J, Lee SJ, Lightfoot M, Milburn N, Mosafer J, Moses A, Murphy DA, Nielsen K, Ocasio MA, Polanco D, Ramos W, Reback CJ, Rezvan PH, Rotheram-Borus MJ, Tang W, Tapia Y, Thomas D, Urauchi S. Online Peer Support for Youth at Higher Risk of or Living with HIV: A Qualitative Content Analysis. AIDS Behav. 2025 Jul;29(7):2135-2143. doi: 10.1007/s10461-025-04677-z. Epub 2025 Mar 16. PMID 40089955
- [Derived] Swendeman D, Rotheram-Borus MJ, Arnold EM, Fernandez MI, Comulada WS, Lee SJ, Ocasio MA, Ishimoto K, Gertsch W, Duan N, Reback CJ, Murphy DA, Lewis KA; Adolescent HIV Medicine Trials Network (ATN) CARES Study Team. Optimal strategies to improve uptake of and adherence to HIV prevention among young people at risk for HIV acquisition in the USA (ATN 149): a randomised, controlled, factorial trial. Lancet Digit Health. 2024 Mar;6(3):e187-e200. doi: 10.1016/S2589-7500(23)00252-2. PMID 38395539
- [Derived] Man OM, Ramos WE, Vavala G, Goldbeck C, Ocasio MA, Fournier J, Romero-Espinoza A, Fernandez MI, Swendeman D, Lee SJ, Comulada S, Rotheram-Borus MJ, Klausner JD. Optimizing Screening for Anorectal, Pharyngeal, and Urogenital Chlamydia trachomatis and Neisseria gonorrhoeae Infections in At-Risk Adolescents and Young Adults in New Orleans, Louisiana and Los Angeles, California, United States. Clin Infect Dis. 2021 Nov 2;73(9):e3201-e3209. doi: 10.1093/cid/ciaa1838. PMID 33300564
- [Derived] Swendeman D, Arnold EM, Harris D, Fournier J, Comulada WS, Reback C, Koussa M, Ocasio M, Lee SJ, Kozina L, Fernandez MI, Rotheram MJ; Adolescent Medicine Trials Network (ATN) CARES Team. Text-Messaging, Online Peer Support Group, and Coaching Strategies to Optimize the HIV Prevention Continuum for Youth: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Aug 9;8(8):e11165. doi: 10.2196/11165. PMID 31400109
- [Derived] Shannon CL, Koussa M, Lee SJ, Fournier J, Abdalian SE, Rotheram MJ, Klausner JD; Adolescent Medicine Trials Network CARES Team. Community-Based, Point-of-Care Sexually Transmitted Infection Screening Among High-Risk Adolescents in Los Angeles and New Orleans: Protocol for a Mixed-Methods Study. JMIR Res Protoc. 2019 Mar 22;8(3):e10795. doi: 10.2196/10795. PMID 30900994
- See also: Annual HIV surveillance report. (2013). LADPH. — http://publichealth.lacounty.gov/wwwfiles/ph/hae/hiv/2013AnnualSurveillanceReport.pdf
- See also: NIH HIV/AIDS Research Priorities and Guidelines for Determining AIDS Funding 2015. — https://grants.nih.gov/grants/guide/notice-files/NOT-OD-15-137.html
- See also: Teens, Social Media & Technology Overview. (2015). Lenhart, A. — http://www.pewinternet.org/2015/04/09/teens-social-media-technology-2015/